CLINICAL TRIAL REGISTRATION COVER PAGE 6-17-21

**RECORD OWNER: JSimmons** 

TITLE: OPIOIDS AND POLICE SAFETY STUDY

DOCUMENT: CONSENT FORM (in PDF/A format)

NCT: not yet provided



Janie Simmons, Ed.D.

Principal Investigator



Department of Social & Behavioral Sciences School of Global Public Health New York University 665 Broadway, 11th Floor, Room 1130 New York, NY 10012

P: 212 992 3807 janies@nyu.edu

# Consent Form

(Study Number: IRB-FY2019-3315)

You are invited to participate in this research study called "Opioids and Police Safety."
This consent form describes the research study, what you may expect if you decide to take part, and important information to help you make your decision.

Please read this form carefully.

#### Why is this study being done?

The purpose of this research project is to develop a successful training for law enforcement officers to equip officers with knowledge and best practices for minimizing workplace harms related to encounters with people who use opioids and/or inject drugs. The Principal Investigator who leads the study is Dr. Janie Simmons. She is an Associate Research Scientist in the School of Global Public Health at New York University. The study will take place online with police officers from Pennsylvania.

### What will I be asked to do if I agree to take part in this study?

If you decide to participate, you will be asked to complete two online trainings, and a series (5) of online surveys over a one-year period. In addition, some officers will also be asked to participate in a brief online interview.

#### Here are the details:

- Follow the instructions in the OPS flyer (enclosed) to enroll in the study.
- Complete an online questionnaire about your background and your experiences with opioid overdoses, people who use drugs, and COVID-19.
- Complete two online trainings -- one on responding to opioid overdoses and the other on minimizing workplace harms. (You will also need to answer a few questions before and after taking the training to assess what you have learned).
- Over the next year, you will complete four brief follow-up surveys (once every 3 months) about your perspectives on the opioid epidemic and your experiences responding to overdoses and people who use drugs. Surveys may also include questions about COVID-19 (including how to prevent its spread and what you think about current responses to this pandemic).

 Some officers (about 30) will be selected at random to take part in a recorded, confidential Zoom or telephone interview with a member of the research team to answer questions about their individual experiences and perspectives.

#### How long will this study take?

Our research team has worked to keep the length of this study as brief as possible. Participation in this study will involve:

- Approximately 30 minutes to enroll in the study and complete the initial online survey.
- Approximately 45-60 minutes to complete each online training.
- Approximately 30 minutes to complete each quarterly follow-up survey.
- If you are selected to be interviewed, approximately 45 minutes to complete your Zoom or telephone interview.

## What possible risks or discomforts can I expect?

This is a minimal risk study, which means that any harms or discomforts that you might experience as a research participant are not any greater than what you would ordinarily encounter in daily life. However, there are some risks to consider:

- The primary risk is that the topic of witnessing or responding to events associated with overdoses or COVID-19 may be upsetting. As a result, you may feel uncomfortable answering survey or interview questions. Questions could provoke sadness, remorse or other emotions.
- There may be a risk to the confidentiality of your data. This means that it may be
  possible to link your survey responses back to you. However, extensive efforts will be
  made to protect your confidentiality and your data. All of your responses to each survey
  and interview will be stored by code number, not by name or other potentially identifying
  information. We will also report all survey data at the group-level and never individually.

(Please also see "Methods to Protect Confidentiality" below on this consent form to learn more.)

#### Will I be compensated for my time?

- Yes! As soon as you enroll, complete the trainings, and the two initial surveys (one before the training; one after the training), you will receive \$75 dollars on your gift card.
- You will receive an additional \$40 on your gift card each time you participate in a follow up survey (total amount of funds possible after initial training and completion of each follow up questionnaire = \$235).
- If you are randomly selected for a telephone interview, an additional \$50 will be added to your gift card (CT card).

#### What possible benefits can I expect from taking part in this study?

You may benefit from participating in this study in the following ways:

- You may benefit by feeling more confident and competent to intervene in overdose emergencies.
- You may benefit from feeling more capable of addressing other potential impacts of the overdose crisis (e.g. preventing needlestick injuries, fentanyl exposure, and burnout).
- You may benefit from being better able to manage psychological risks and stressors when responding to overdose events and COVID-19 (i.e. self-care practices, encouraging help-seeking behavior, providing resource lists.
- You may benefit from learning how to mitigate risks associated with COVID-19.

#### Methods to Protect Confidentiality

Our research team will work carefully to ensure confidentiality of your personal data (your name, email, phone number, data collected) by doing the following:

- You will be assigned a unique identification (ID) number that will be used (instead of your name) on all enrollment forms, questionnaires, surveys, interviews, transcripts and other research materials.
- The online data collection website that our study will be using does not collect any identifying information. Only your unique ID number will be used.
- Only this signed consent form will link your name to your ID number. The locator form
  that our research team needs to help keep track of your data will not contain the
  participant's ID numbers and will be kept in a separate locked file cabinet at New York
  University and in a secure password-protected, encrypted, computer file.
- Interview data (stored as audio and video files) will be secured on a secure, password
  protected, encrypted computer file. Once the audio file is transcribed, the video portion of
  the recording will be deleted (destroyed).
- Information that does *not* contain your personal information may be used in future research, shared with other researchers, and/or placed in a data repository without your additional consent.
- The study will be registered at clinicaltrials.gov and some information may be posted, including demographic and baseline characteristics, outcomes and statistical analyses, any adverse events, though identifiers, such as name and contact info will remain confidential.

#### When is the study over? Can I leave before it ends?

The study is over when you have completed the last follow-up survey. Participation in this study is voluntary. You may refuse to participate or withdraw at any time without penalty. For interviews or surveys, you have the right to skip or refuse to answer any questions you prefer not to answer.

#### **Additional Information**

If there is anything about the study or your participation that is unclear or that you do not understand, or if you have questions or wish to report a research-related problem, you may contact Dr. Janie Simmons at (212) 992-3807 or js8822@nyu.edu, 665 Broadway, Room 1130. For questions about your rights as a research participant, you may contact the University Committee on Activities Involving Human Subjects (UCAIHS), New York University, 665 Broadway, Suite 804, New York, New York, 10012, at ask.humansubjects@nyu.edu or (212) 998-4808. Please reference the study # (IRB-FY2019-3315) when contacting the IRB (UCAIHS). Once you have completed this consent form, save it as a pdf and print it or store it on your computer so you have a copy.

| Agreement to Participate |
|--------------------------|
| Your Signature & Date |